CLINICAL TRIAL: NCT00568438
Title: Immunohistochemical & Immunoblot Analysis of NIS (Na+/I-Symporter) in Archival and Frozen Human Tissue Samples
Brief Title: Immunohistochemical & Immunoblot Analysis of NIS (Na+/I-Symporter) in Archival & Frozen Tissue Sample
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-11005; BRSNSTU0011 (Other: OnCore)
Record Dates: First submitted 2007-12-04; First posted 2007-12-06 (Estimated); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Breast Cancer; Stomach Neoplasms; Salivary Gland Neoplasms; Thyroid Cancer
MeSH Terms: conditions — Breast Neoplasms; Stomach Neoplasms; Salivary Gland Neoplasms; Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Cases will be identified from clinic patient medical records and linked to pathology reports. The surgical pathology record number will thus be obtained and used to retrieve the archival blocks and slides. Approximately three representative blocks will be selected and 4-6 four micron thick sections will be cut on a microtome. Cases with limited archived diagnostic material will not be selected nor blocks where there is little materials.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this study is to study NIS expression in benign and malignant breast and thyroid samples using archival formalin-fixed paraffin-embedded tissue sections.

DETAILED DESCRIPTION:
The objective of the study is to further understanding of proteins that occur in both normal cells and tumor cells and to learn more about certain diseases and potential alternative treatments for these diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be over the age of 18.
2. Patients must have benign and malignant breast and thyroid cancer.
3. Patient mus sign consent form.

Exclusion Criteria:

1. No children will be allowed.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cases will be identified from clinic patient medical records and linked to pathology reports. The surgical pathology record number will thus be obtained and used to retrieve the archival blocks and slides. In addition, all these participants will be clinical patients of the Protocol Director, thus the Physician will always be familiar with the participants.
Sampling Method: Non-Probability Sample
Enrollment: 169 (Actual)
Dates: Start 2000-10; Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irene L Wapnir, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No